CLINICAL TRIAL: NCT06562140
Title: Multidimensional Examination of Physical Activity, Functional Capacity, and Health Status in Patients with Colorectal and Anal Cancer
Brief Title: Multidimensional Examination of Patients with Colorectal and Anal Cancer
Acronym: MECACP
Status: Recruiting | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Alexandra Makai, senior lecturer, University of Pecs
Other Study IDs: 9636-PTE-2023
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer; Anal Cancer; Physical Inactivity; Fecal Incontinence; Quality of Life
Keywords: colorectal cancer; anal cancer; quality of life; physical activity; fecal incontinence
MeSH Terms: conditions — Colorectal Neoplasms; Anus Neoplasms; Sedentary Behavior; Fecal Incontinence; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Colorectal cancer patients: Patients aged 18 to 80 years with a diagnosis of colorectal carcinoma
  Interventions: Other: No intervention - cross-sectional observational study
- Anal cancer patients: Patients aged 18 to 80 years with a diagnosis of anal carcinoma
  Interventions: Other: No intervention - cross-sectional observational study

INTERVENTIONS:
Other: No intervention - cross-sectional observational study — No intervention - cross-sectional observational study

SUMMARY:
The aim of our cross-sectional research is to assess changes in physical activity, functional capacity, and health status in individuals with colorectal and anal carcinoma using subjective measurement tools, with particular focus on those suffering from incontinence, through a cross-sectional study. Additionally, the research involves the Hungarian adaptation and validation of the quality of life questionnaire for colorectal cancer (EORTC QLQ-CR29), quality of life questionnaire for anal cancer (EORTC QLQ-AN27), and Fecal Incontinence Severity Index (FISI)" questionnaires.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most commonly diagnosed cancer and the second leading cause of cancer-related deaths worldwide. The incidence of CRC is known to be high in developed countries and increases with socioeconomic development. Well-known risk factors include aging, alcohol consumption, smoking, and obesity. In addition to family history, lifestyle changes in diet, occupation, or physical activity may also emerge as risk factors for CRC. Previous research findings have shown a significant association between reduced physical activity and an increased risk of CRC. With improved patient survival rates, functional outcomes such as fecal incontinence, urinary, and sexual dysfunction are becoming increasingly important, as they are known to significantly impact quality of life (QoL). Reviewing the functional outcomes of rectal cancer surgeries, it is observed that even years after surgery, one-third of patients suffer from fecal incontinence. In contrast, studies on the functional outcomes following colon cancer surgeries are rare and often involve relatively small study populations. Previous studies have shown that physical activity in cancer survivors can have numerous beneficial health effects and is associated with a reduced risk of cancer recurrence and mortality in cases of colon and rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* adult (18-80 years) patients with a diagnosis of colorectal or anal carcinoma

Exclusion Criteria:

* Neuromuscular diseases
* severe congenital musculoskeletal and other disorders,
* severe psychiatric illness, lack of cooperation,
* undergone other surgical procedures within the past year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is colorectal or anal cancer patients older than 18 years. Neuromuscular diseases, severe congenital musculoskeletal and other disorders, severe psychiatric illness, lack of cooperation, undergone other surgical procedures within the past year.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life questionnaire for cancer patients - EORTC QLQ-C30 | Baseline
  The EORTC QLQ-C30 questionnaire examines the general impact of cancer and its treatment. The minimum value is 30, maximum 120, where higher scores means worse health-related quality of life.
Quality of life questionnaire for colorectal cancer - EORTC QLQ-CR29 | Baseline
  The EORTC QLQ-CR29 questionnaire assesses the general impact of cancer and its treatment among colorectal cancer patients. The minimum value is 29, maximum 116, where higher scores means worse health-related quality of life
Quality of life questionnaire for anal cancer - EORTC QLQ-AN27 | Baseline
  The EORTC QLQ-CR29 questionnaire assesses the general impact of cancer and its treatment among anal cancer patients. The minimum value is 27, maximum 108, where higher scores means worse health-related quality of life
Global Physical Activity Questionnaire (GPAQ) | 1 week
  To measure physical activity patterns related to work, active transportation, leisure time activities and sitting time. The work time physical activity, active transportation, recreational activities and sitting time will be summarized as weekly minutes.
FECAL INCONTINENCE SEVERITY INDEX (FISI) | Baseline
  The questionnaire measures the frequency of the different incontinence events and the type of stool involved. The index provides a numerical score that reflects the overall severity of a patient's fecal incontinence. A total score is the sum of all points between 0 to 61, where the higher the score means more severe fecal incontinence.

CONTACTS AND LOCATIONS:
Locations (2):
- Hungary (2):
  - University of Pécs, Pécs, Baranya
  - University of Pécs, Pécs

IPD SHARING:
Plan to Share IPD: Undecided